CLINICAL TRIAL: NCT03605316
Title: Electric Neuromodulation in Refractory Obsessive-compulsive Disorder : the Montpellier Experience (France)
Brief Title: Deep Electrical Neuromodulation in Obsessive-compulsive Disorder
Acronym: NEP-TOC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0141
Record Dates: First submitted 2018-04-13; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-04

CONDITIONS: Obsessive-compulsive Disorder (OCD)
Keywords: Deep brain stimulation; obsessive-compulsive disorder; neuromodulation; psychiatry; quality of life
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Deep brain stimulation (DBS) — Neurosurgical treatment by stereotactic implantation of electrodes in the brain that affects the functioning of subcortical neuronal circuits

SUMMARY:
Obsessive-compulsive disorder (OCD) is a neuropsychiatric disease characterised by intrusive, recurrent and persistent thoughts, urges or images (obsessions) and the resulting excessive repetitive behaviours or mental acts according to rigid rules unrealistically aimed at reducing distress (compulsions).

Its lifetime prevalence in the general population is usually estimated between 1 - 3% (Ruscio, Mol Psychiatry, 2010). Despite appropriate pharmacological and cognitive-behavioural treatments, it is commonly estimated that 10% of patients are therapy-refractory and that among improved or recovered patients, sustained efficacy is uncertain.

For treatment refractory OCD patients, a neurosurgical treatment by deep brain stimulation (DBS), has emerged in the late 1990s as a new therapeutic option (Nuttin et al, Lancet, 1999).

The objective of the current study is to report the long-term treatment effects (safety and effectiveness) of DBS from the cohort of six severe and therapy-refractory OCD patients implanted at the French university hospital of Montpellier since 2003.

DETAILED DESCRIPTION:
The data needed to carry out the study will be extracted from the medical files of the 6 patients concerned.

The following data will be collected:

* Age, sex
* Medical, surgical and psychiatric history
* History of pharmacological treatments
* Elements from clinical examination
* any reported adverse effect
* scores of the various questionnaires completed throughout the follow-up (including Y-BOCS and GAF)
* results of biological, morphological, neuropsychological tests
* Stimulation parameters applied since implantation.

ELIGIBILITY:
Inclusion criteria:

* all patients with severe and refractory OCD according to DSM-IV criteria, confirmed by experienced psychiatrist
* treated by DBS at the CHU of Montpellier

Exclusion criteria:

- already enrolled in a study protocol at time of implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Six patients consisting in three males and three females aged 18 years and over implanted at the University Hospital (CHU) of Montpellier (France) between June 2003 and February 2013.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline
  10-item scale with scores ranging from 0 to 40; higher scores indicating more severe OCD symptoms.
  Patients are defined as responders if they have a score decrease of at least 35% on the Y-BOCS
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 12 months
  10-item scale with scores ranging from 0 to 40; higher scores indicating more severe OCD symptoms.
  Patients are defined as responders if they have a score decrease of at least 35% on the Y-BOCS

SECONDARY OUTCOMES:
Global Assessment of Functioning (GAF), axis V of the DSM-IV (APA, 1994). | Baseline
  a rating scale used to subjectively assess the social and occupational functioning as well as psychological symptoms of adults. The scale ranges from 1 to 100, divided into 10-point intervals describing the level of functioning and symptoms.
Global Assessment of Functioning (GAF), axis V of the DSM-IV (APA, 1994). | 12 months
  a rating scale used to subjectively assess the social and occupational functioning as well as psychological symptoms of adults. The scale ranges from 1 to 100, divided into 10-point intervals describing the level of functioning and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne CYPRIEN, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC